CLINICAL TRIAL: NCT01575119
Title: Decision Aid Development for Cigarette Smokers Undergoing Surgery: Specific Aim 2
Brief Title: Decision Aid for Cigarette Smokers Undergoing Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Warner, Associate Director of Clinical and Translational Research, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-009150
Record Dates: First submitted 2012-04-05; First posted 2012-04-11 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Tobacco Abuse
Keywords: Cigarette smoker; Elective surgery
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- In-patient surgery (Experimental): Decision Aid tool is presented by respiratory therapist, prompting a discussion with the provider (physician or physician assistant)about smoking around time of surgery
  Interventions: Behavioral: Decision Aid
- In-patient (Active Comparator): Standard of care information, including distributing patient education brochure, to provide information regarding perioperative smoking
  Interventions: Behavioral: Control intervention
- Out-patient surgery (Experimental): Decision Aid tool is presented by respiratory therapist, prompting a discussion with the provider (physician or physician assistant)about smoking around time of surgery
  Interventions: Behavioral: Decision Aid
- Out-patient (Active Comparator): Standard of care information, including distributing a patient education brochure, to provide information regarding perioperative smoking
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Decision Aid — Decision Aid tool is presented by respiratory therapist, prompting a discussion with the provider (physician or physician assistant)about smoking around time of surgery
  Arms: In-patient surgery
Behavioral: Control intervention — Standard of care information, including distributing patent education brochure, to provide information regarding perioperative smoking
  Arms: In-patient
Behavioral: Decision Aid — Decision Aid tool is presented by respiratory therapist, prompting a discussion with the provider (physician or physician assistant)about smoking around time of surgery
  Arms: Out-patient surgery
Behavioral: Control — Standard of care information, including distributing patient education brochure, to provide information regarding perioperative smoking
  Arms: Out-patient

SUMMARY:
Smokers have three choices when faced with surgery: keep smoking, quit for a short time around surgery or quit for good. In the first specific aim, a decision aid was designed to help facilitate the discussion of these choices between smokers and healthcare providers. This second aim will test whether this decision aid improves the decisional quality compared with standard methods used to discuss perioperative smoking.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker
* Scheduled to undergo elective surgery at Mayo Clinic Rochester
* Age 18 years or older
* Able to fully participate in all study aspects

Exclusion Criteria:

* Unavailable for telephone follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Measures of decisional quality | Assessed immediately after the time of the preoperative conversation in the preoperative clinic
  The Decisional Conflict Scale and the OPTION Scale will be utilized

SECONDARY OUTCOMES:
Measures of intent and self-efficacy | Immediately after the preoperative evaluation in the preoperative clinic
  Intent to quit smoking, and self-efficacy for quitting

CONTACTS AND LOCATIONS:
Overall Officials: David Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States